CLINICAL TRIAL: NCT02919345
Title: Comparative Study of Dapagliflozin Versus Glibenclamide Effect on Endothelial Function of Coronary Artery Disease Patients
Brief Title: Assessment of Dapagliflozin Effect on Diabetic Endothelial Dysfunction of Brachial Artery
Acronym: ADDENDA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, MD, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Artery Disease; Carotid Artery Diseases
Keywords: Dapagliflozin; Glibenclamide; Endothelial Function; Vascular Endothelial Cells; Flow Mediated Dilation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Carotid Artery Diseases | interventions — dapagliflozin; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg in addition to Metformin 1500 mg
  Interventions: Drug: Dapagliflozin 10 mg
- Glibenclamide (Active Comparator): Glibenclamide 5mg in addition to Metformin 1500 mg
  Interventions: Drug: Glibenclamide 5 mg

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — Dapagliflozin 10 mg in addition to Metformin 1500 mg/day
  Other Names: Farxiga
  Arms: Dapagliflozin
Drug: Glibenclamide 5 mg — Glibenclamide 5 mg in addition to Metformin 1500 mg/day
  Other Names: Daonil, Glyburide
  Arms: Glibenclamide

SUMMARY:
Background Endothelial dysfunction is one of the early events in atherosclerotic plaque development. It is characterized by an increased ratio of substances with vasoconstrictive, pro-thrombotic, and proliferative properties over substances with vasolidatory, antithrombogenic and antimitogenic properties. Endothelial dysfunction is also associated with high-risk patients with coronary artery disease. Hyperglycemia, obesity, hypertension and fat mass also impair the endothelium by increasing the expression of cytokines, inflammatory markers and vascular markers.

Hypothesis Administration of dapagliflozin in addition to metformin background with clinical or subclinical cardiovascular atherosclerotic disease improves endothelial function when compared to those using glibenclamide in addition to metformin.

Objectives Evaluate the effect of dapagliflozin vs glibenclamide on a metformin background on endothelial function in patients with clinical or subclinical cardiovascular atherosclerotic disease and poorly controlled diabetes.

Enpoints Prymary Change in flow mediated dilation (FMD) and its related endpoint (FMD post reperfusion lesion) between the randomization visit and over 12 weeks of treatment.

Secondary Change in plasma nitric oxide, isoprostane, ICAM-1, VCAM-1, ET-1, leptin, adiponectin, C-reactive protein, TNF- α, interleukin-6, interleukin-2, weight and body composition (% of fat mass and % free fat mass) at the randomization visit and over 12 weeks of treatment.

3

Design Randomized, parallel-group, comparative, prospective clinical study. The study is divided in two phases: Run-in and Randomization. In the former phase, which must have the maximum period of 16 weeks, patients will visit the outpatient to adjust metformin and blood pressure medications. After run-in phase, patients that fulfill inclusion criteria will perform an ambulatory blood pressure monitoring (ABPM) in order to asses BP; body composition will be assessed by dual x-ray absorptiometry (DXA); endothelial function as assessed by flow mediated dilation and vascular cytokines. Patients will by randomized to dapagliflozin or glibenclamide on a metformin background. After 12 weeks, the ABPM, DXA and endothelial function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

(i) chronic coronary artery disease as shown by angiogram or subclinical artery disease diagnosed by the presence of carotid atherosclerotic plaque or carotid Intima-Media Thickness (cIMT) ≥ 1mm;

(ii) T2DM using up to two oral hypoglycemic agents;

(iii) inadequate glycemic control (HbA1c ≥ 7%);

Exclusion Criteria:

(i) HbA1c > 9%;

(ii) contraindications to metformin use (Cr Clearance <60 ml/min, Cr> 1.5 mg/dL in men and> 1.4 mg/dl in women, liver failure - AST or ALT> 3x upper normal limit or other conditions that might increase the risk of lactic acidosis);

(vi) at the time of randomization, patient who is not on metformin XR 1500 mg/day monotherapy for at least 12 weeks;

(vii) patients who spend more than 16 weeks to adjust metformin before randomization;

(viii) BP ≥ 140 x 90 after 16 weeks of anti-hypertensive medication adjustment;

(iii) hospitalization for unstable angina or acute myocardial infarction within 2 months prior to enrolment;

(iv) acute stroke or transient ischemic attack (TIA) within two months prior to enrolment;

(v) less than two months post coronary artery revascularization;

(ix) patients with FMD <2% at the time of randomization;

(x) triglycerides > 500 mg/dL;

(xi) known allergy to any of the study drugs;

(xii) patients with severe coronary artery disease and heart failure;

(xiii) systemic vasculitis;

(xiv) conditions that lead to systemic inflammation;

(xv) patients using rosiglitazone;

(xvi) polyuria, polydipsia, weight loss, or others clinical signs of volume depletion;

(xvii) those who refuse to participate or sign the Statement of Informed Consent;

(xviii) pregnancy or women during reproductive age;

(xix) breastfeeding women;

(xx) history of gastrointestinal disorders that may interfere with the absorption of study medication;

(xxi) patients who are participating in other clinical studies or whose participation ended less than six months ago.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in flow mediated dilation (FMD) and its related endpoint (FMD post reperfusion lesion) | 12 weeks

SECONDARY OUTCOMES:
Change in plasma nitric oxide | 12 weeks
Change in plasma isoprostane | 12 weeks
Change in plasma nitric oxide after reperfusion injury. | 12 weeks
Change in plasma isoprostane after reperfusion injury. | 12 weeks
Change in plasma Intercellular Adhesion Molecule 1(ICAM-1) | 12 weeks
Change in plasma Vascular Cell Adhesion Molecule 1 (VCAM-1) | 12 weeks
Change in plasma Endothelin-1 (ET-1) | 12 weeks
Change in plasma Leptin | 12 weeks
Change in plasma Adiponectin | 12 weeks
Change in plasma C-reactive protein (CRP) | 12 weeks
Change in plasma Tumor Necrosis Factor alpha (TNF-α) | 12 weeks
Change in plasma interleukin-6 | 12 weeks
Change in plasma interleukin-2 | 12 weeks
Change in weight | 12 weeks
Change in body composition (% of fat mass and % free fat mass) | 12 weeks

OTHER OUTCOMES:
Change in Glycated Hemoglobin | 12 weeks
Change in Systolic Blood Pressure | 12 weeks
Change in Mean Arterial Blood Pressure | 12 weeks
Change in Waist Circumference | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- State University of Campinas, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Cintra RMR, Soares AAS, Breder I, Munhoz DB, Barreto J, Kimura-Medorima ST, Cavalcante P, Zanchetta R, Breder JC, Moreira C, Virginio VW, Bonilha I, Lima-Junior JC, Coelho-Filho OR, Wolf VLW, Guerra-Junior G, Oliveira DC, Haeitmann R, Fernandes VHR, Nadruz W, Chaves FRP, Arieta CEL, Quinaglia T, Sposito AC; ADDENDA-BHS2 trial investigators. Assessment of dapagliflozin effect on diabetic endothelial dysfunction of brachial artery (ADDENDA-BHS2 trial): rationale, design, and baseline characteristics of a randomized controlled trial. Diabetol Metab Syndr. 2019 Jul 31;11:62. doi: 10.1186/s13098-019-0457-3. eCollection 2019. PMID 31384310